CLINICAL TRIAL: NCT03815123
Title: Register Kardialer Computertomographie
Status: Recruiting | Type: Observational
Sponsor: Das Radiologische Zentrum (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Principal Investigator, Johannes Görich, Prof. Dr. med. Johannes Görich, Das Radiologische Zentrum
Other Study IDs: S-758/2018
Record Dates: First submitted 2019-01-21; First posted 2019-01-24 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Evaluation of CT in Coronary Artery Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: cardiac CT — The cardiac CT examinations are indicated by the referring physician. The participation in this study has no influence on the further diagnostic and therapeutic regimen.

SUMMARY:
The aim of this Heidelberg Cardiac CT Registry (Register kardiale Computertomographie) is to assess the diagnostic and prognostic perfomance of cardiac CT exminations in a real-world patient population.

DETAILED DESCRIPTION:
Anthropometric data, medical history and results of the CT examinations are collected in a database in order to adressing various scientific questions.

ELIGIBILITY:
Inclusion Criteria:

• Subjects referred for cardiac CT examination by their physician

Exclusion Criteria:

• none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects referred for cardiac CT examination by their physician
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-12-06 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
coronary CT angiography | 10 years
  Evaluation of degree of coronary artery stenosis
coronary CT angiography | 10 years
  Assessment of coronary plaque composition
Agreement with other imaging modalities | 10 years
  Agreement with other imaging modalities
Occurence of MACE | 10 years
  Occurence of major adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Radiologische Praxis Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Andre F, Fortner P, Emami M, Seitz S, Brado M, Guckel F, Sokiranski R, Sommer A, Frey N, Gorich J, Buss SJ. Factors influencing the safety of outpatient coronary CT angiography: a clinical registry study. BMJ Open. 2022 Aug 8;12(8):e058304. doi: 10.1136/bmjopen-2021-058304. PMID 35940836
- See also: Website — https://www.das-radiologische-zentrum.de